CLINICAL TRIAL: NCT02150239
Title: A Survey on Postoperative Pain (POP) Experience in Asian Patients.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Other Study IDs: 20144-137
Record Dates: First submitted 2014-05-26; First posted 2014-05-29 (Estimated); Last update posted 2014-06-10 (Estimated); Status verified 2014-06

CONDITIONS: Postoperative Pain
Keywords: pain; postoperative
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- postoperative pain
  Interventions: Procedure: operation

INTERVENTIONS:
Procedure: operation

SUMMARY:
Pain management is becoming an important ethical responsibility of the medical profession and a focus of the health care system. However, there are limited literature evaluate the postoperative pain experience and management in our local setting.

DETAILED DESCRIPTION:
We need to identify those patients who, from a demographic, psychology and surgical viewpoint, are more at risk of experiencing postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* 1. Adult with age ≥ 18 who undergo operation

Exclusion Criteria:

* 1. Refused to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult with age ≥ 18 who undergo operation
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2014-05; Primary Completion 2014-09 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
postoperative pain experience | 2 weeks
  To determine patient's postoperative pain experience during and 2 weeks after discharge from hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Wang Chew Yin, Principal Investigator — University of Malaya
Locations (1):
- University Malaya Medical Center, Kuala Lumpur, KL, Malaysia